CLINICAL TRIAL: NCT01463189
Title: Web-based Support to Manage Arthritis Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Inflexxion, Inc. (Industry)
Responsible Party: Principal Investigator, Kimberlee Trudeau, Research Scientist, Inflexxion, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5R44AR061191 (NIH)
Record Dates: First submitted 2011-10-20; First posted 2011-11-01 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Ankylosing Spondylitis; Other Arthritic Conditions (e.g., Psoriatic Arthritis)
Keywords: arthritis; self management
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic; Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- painACTION: Arthritis (Experimental)
  Interventions: Behavioral: painACTION: Arthritis
- treatment as usual (No Intervention)

INTERVENTIONS:
Behavioral: painACTION: Arthritis — Participants will be asked to complete eight 20-minute sessions on the site over a four-week intervention period (two site visits per week), and complete five 20-minute "booster" sessions (one site visit per month) during the follow up period. Each session will have a minimum set of requirements. Specific details about the requirements for each session will be provided in the session logs.
  Arms: painACTION: Arthritis

SUMMARY:
Development of an interactive, online pain self-management program for adults who suffer from pain associated with osteoarthritis, rheumatoid arthritis, Ankylosing spondylitis, and other arthritic conditions (e.g., psoriatic arthritis) using principles from Social Cognitive Theory (Bandura, 1977). This online health intervention, painACTION: Arthritis, will provide clinically reliable information about diagnosis, treatment, and management of arthritis, written for health consumers in a clear and engaging manner to help increase their skills and confidence to use self-management strategies.

DETAILED DESCRIPTION:
One of every five adults in the United States (46.4 million people) is affected by arthritis. Increasing the number of days individuals are free of arthritis pain is one of the Healthy People 2010 objectives. Although there are a variety of medical treatments and medications available, self-management is a critical component in helping arthritis sufferers learn how to identify, avoid, and help manage their pain. Unfortunately, clinicians face significant time pressure, leaving little time for desired patient-provider education and collaboration. This is an important omission as tailored advice (e.g., specific exercises to reduce pain) from health providers could enable behavior change and improve outcomes. Therefore, widely accessible and tailored interventions that address motivational issues are needed to facilitate self-management education among arthritis patients. Because of its reach across demographic groups, the Internet is an excellent vehicle for offering a self-management program to arthritis sufferers. The investigators propose to develop an interactive, online pain self-management program for adults who suffer from pain associated with osteoarthritis, rheumatoid arthritis, Ankylosing spondylitis, and other arthritic conditions (e.g., psoriatic arthritis) using principles from Social Cognitive Theory (Bandura, 1977). This online health intervention, painACTION: Arthritis, will provide clinically reliable information about diagnosis, treatment, and management of arthritis, written for health consumers in a clear and engaging manner to help increase their skills and confidence to use self-management strategies. Moreover, it will be designed to complement and connect to our other SBIR-supported pain online health interventions (chronic back pain, migraine pain, neuropathic pain) to be a more comprehensive resource for those seeking pain management assistance. The most unique aspect of painACTION: Arthritis is that it includes three technological innovations -- a Web 2.0-enabled platform, a Custom Recommendation Engine, and Dynamic Lessons - to help people self manage their arthritis pain. In Phase I the investigators accomplished two important objectives: 1) established the feasibility of painACTION: Arthritis as an intervention and a technical project and 2) generated preliminary plans for the content, design, and technical development of painACTION: Arthritis. In Phase II the investigators will produce the program and test its efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age;
2. Be able to provide informed consent
3. Be able to read and speak English
4. Have reliable Internet access and e-mail
5. Have a self-reported doctor diagnosis of arthritis, limited to the following conditions - osteoarthritis (OA), rheumatoid arthritis (RA), ankylosing spondylitis (AS), or other arthritis conditions (e.g., psoriatic arthritis)
6. Have a self-reported pain level of 4 or more in the past week on the 0 to 10 Numeric Rating Scale (McCaffery & Beebe, 1993) because 4 indicates moderate or higher level of pain.

Exclusion Criteria:

1. Participation in another Inflexxion pain management study.
2. Participation in an online research study related to arthritis in the past year
3. Currently in pain from a recent injury
4. Has been hospitalized for non-medical reasons related to emotional or mental health in the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2011-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change in cognitions from baseline to: post intervention (approximately 1 month post baseline), 3 months post intervention, 6 months post intervention | baseline, post intervention, 3 months post intervention, and 6 months post intervention
  Arthritis Self-efficacy Scale (Lorig et al., 1989) is an 8-item questionnaire that assesses a patient's ability to determine self-efficacy.
  Pain Catastrophizing Scale (PCS) (Sullivan et al., 1995) was developed to assess three components of catastrophizing: rumination, magnification, and helplessness. The scale consists of 13 items rated from 0-4 (0 = not at all, 4 = all the time).
  Pain Awareness Questionnaire (Berman et al., 2009) is a 7-item questionnaire that assesses a patient's awareness of their current pain.
Change in self management behaviors from baseline to: post intervention post intervention (approximately 1 month post baseline), 3 months post intervention, 6 months post intervention | baseline, post-intervention, 3 months post-intervention, and 6 months post-intervention
  Exercise Behaviors (Lorig et al., 1996) is a 6-item questionnaire assessing the total time a patient had participated in various forms of exercise (e.g., stretching).
  Cognitive Symptom Management (Lorig et al., 1996) is a 6-item questionnaire assessing a patient's ability to manage their symptoms. This scale is rated on a 0 to 5 scale: 0 = never to 5 = always.
  Communication with Physicians (Lorig et al., 1996) is a 3-item scale assessing a patient's communication with their physicians. This scale is rated on a 0 to 5 scale: 0 = never to 5 = always.
Change in pain and functioning from baseline to: post intervention post intervention (approximately 1 month post baseline), 3 months post intervention, 6 months post intervention | baseline, post-intervention, 3 months post-intervention, and 6 months post-intervention
  Brief Pain Inventory - Short Form (BPI-SF) (Cleeland, 1991) uses a 0 to 10 numeric rating scale to obtain information on the intensity of pain, the degree to which pain interferes with function, pain relief, pain quality, and the patient's perception of the cause of pain (6 items).

SECONDARY OUTCOMES:
Change in quality of life from baseline to: post intervention post intervention (approximately 1 month post baseline), 3 months post intervention, 6 months post intervention | baseline, post intervention, 3 months post intervention, and 6 months post intervention
  The Arthritis Impact Measurement Scale-2-SF (Guillemin et al., 1997) is a 26-item scale that measures 5-domains of health status (e.g., physical, role, work, and social functioning.) Six additional items from the Ankylosing Spondylitis-AIMS will be added for additional validity of spine and mobility functioning for the participants with AS (Guillemin et al., 1999).
  Patient Global Impression of Change Scale (Guy, 1976) is an outcome measure of global improvement with treatment and consists of a single-item self-rating.
Change in affect from baseline to: post intervention post intervention (approximately 1 month post baseline), 3 months post intervention, 6 months post intervention | baseline, post-intervention, 3 months post-intervention, and 6 months post-intervention
  Depression Anxiety Stress Scales (DASS-21, Lovibond & Lovibond, 1995). The DASS is a 21-item questionnaire that distinguishes symptoms of depression, anxiety, and stress.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberlee J Trudeau, Ph.D., Principal Investigator — Inflexxion, Inc.
Locations (1):
- Inflexxion, Inc., Newton, Massachusetts, United States

REFERENCES:
- [Background] Bandura A. Self-efficacy: toward a unifying theory of behavioral change. Psychol Rev. 1977 Mar;84(2):191-215. doi: 10.1037//0033-295x.84.2.191. No abstract available. PMID 847061
- [Background] Lorig K, Chastain RL, Ung E, Shoor S, Holman HR. Development and evaluation of a scale to measure perceived self-efficacy in people with arthritis. Arthritis Rheum. 1989 Jan;32(1):37-44. doi: 10.1002/anr.1780320107. PMID 2912463
- [Background] Lorig K, Stewart A, Ritter P, González V, Laurent D, Lynch J. Outcome measures for health education and other health care interventions. Thousand Oaks, CA: Sage Publications, 1996.
- [Background] Sullivan MJL. The pain catastrophizing scale: Development and validation. Psychological Assessment 7(4):524-532, 1995.
- [Background] Berman RL, Iris MA, Bode R, Drengenberg C. The effectiveness of an online mind-body intervention for older adults with chronic pain. J Pain. 2009 Jan;10(1):68-79. doi: 10.1016/j.jpain.2008.07.006. Epub 2008 Sep 5. PMID 18774342
- [Background] Cleeland CS. Brief Pain Inventory (Short Form). Pain Research Group. Retrieved March 17, 2009, from http://prc.coh.org/pdf/BPI%20Short%20Version.pdf, 1991.
- [Background] Guillemin F, Coste J, Pouchot J, Ghezail M, Bregeon C, Sany J. The AIMS2-SF: a short form of the Arthritis Impact Measurement Scales 2. French Quality of Life in Rheumatology Group. Arthritis Rheum. 1997 Jul;40(7):1267-74. doi: 10.1002/1529-0131(199707)40:73.0.CO;2-L. PMID 9214427
- [Background] Guillemin F, Challier B, Urlacher F, Vancon G, Pourel J. Quality of life in ankylosing spondylitis: validation of the ankylosing spondylitis Arthritis Impact Measurement Scales 2, a modified Arthritis Impact Measurement Scales Questionnaire. Arthritis Care Res. 1999 Jun;12(3):157-62. doi: 10.1002/1529-0131(199906)12:33.0.co;2-r. PMID 10513505
- [Background] Guy W. ECDEU Assessment Manual for Psychopharmacology. Rockville, MD: U.S. Department of Health, Education, and Welfare, 1976.
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] McCaffery M, Beebe A. Pain: Clinical Manual for Nursing Practice. Baltimore: V.V. Mosby Company, 1993.